CLINICAL TRIAL: NCT03656198
Title: Non-specific Effects of Rabies Vaccine on the Incidence of Common Infectious Disease Episodes: a Randomized Controlled Trial
Brief Title: Non-specific Effects of Rabies Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ross University School of Veterinary Medicine (Other)
Collaborators: Serum Institute of India Pvt. Ltd. (Industry)
Responsible Party: Principal Investigator, Darryn Knobel, Professor of Epidemiology and Population Health, Ross University School of Veterinary Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 18-04-FL
Record Dates: First submitted 2018-08-24; First posted 2018-09-04 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Influenza-like Illness; Upper Respiratory Disease; Diarrhea; Fever
Keywords: Non-Specific Effects of Vaccines; Heterologous Immunity; Rabies; Patient Reported Outcome Measures
MeSH Terms: conditions — Respiration Disorders; Diarrhea; Fever; Rabies

STUDY DESIGN:
Intervention Model Description: The trial design is a single-site, two-arm, parallel-group, participant-blinded, randomized, placebo-controlled, two-sided comparative study, with an internal pilot study for blinded sample size re-estimation. Allocation to study arm will be by block randomization stratified by sex within cohort (semester) with a 1:1 allocation ratio.
Who Masked: Participant
Masking Description: Participants will be blinded to their study arm allocation. The intervention procedure will be identical for both arms (intramuscular injections at Student Health Services on days 0, 7 and 21). Participants allocated to the control group will receive an intramuscular injection of sterile water for injection using identical syringes and needles as for the vaccine group. The injection will be prepared in a separate room to maintain participant blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaccine group (Experimental): Three dose primary course of Rabivax-S. Dosing and administration of the vaccine (Rabivax-S) will be according to the package insert, following the schedule for pre-exposure prophylaxis via the intramuscular route; that is, 1 mL by intramuscular injection in the deltoid area of the arm on Day 0, Day 7 and Day 21.
  Interventions: Biological: Rabivax-S
- Control group (Placebo Comparator): The intervention (placebo) in the control group is at least one dose (1 mL by intramuscular injection) of a three dose primary course (on days 0, 7 and 21) of vaccine diluent (sterile water for injection).
  Interventions: Drug: Sterile Water Injection

INTERVENTIONS:
Biological: Rabivax-S — Rabivax-S is a lyophilized vaccine manufactured by Serum Institute of India Pvt. Ltd. containing inactivated purified rabies antigen (Pitman Moore, PM3218 as virus strain) produced using Vero ATCC CCL 81 cells. The diluent (sterile water for injection) is provided in a separate 1 mL ampoule. After reconstitution, a single dose of 1 mL contains an inactivated, purified rabies antigen (not less than 2.5 IU), glycine (40 mg), sucrose (40 mg) and human serum albumin (25% 10 mg).
  Arms: Vaccine group
Drug: Sterile Water Injection — The vaccine diluent (sterile water for injection) is provided in a separate 1 mL ampoule.
  Arms: Control group

SUMMARY:
Vaccines work by stimulating the body to produce a high-quality, rapid and specific immune response upon exposure to infection by a particular disease-causing microorganism - the microorganism targeted by the vaccine. Evidence is emerging that some vaccines may have additional 'non-specific effects' (NSEs); that is, effects on the immune system beyond the direct protection against the diseases for which the vaccines were developed. It has been proposed that rabies vaccine has protective NSEs in people and animals, with receipt of rabies vaccine in children associated with a reduced risk of meningitis and cerebral malaria in one study, and a history of rabies vaccination in free-roaming dogs associated with increased survival rates in another study. Studies in mice have shown that prior rabies vaccination protects against bacterial sepsis. The biological mechanism of action of any such NSE of rabies vaccine is unknown. Other vaccines with reported protective NSEs (e.g. bacillus Calmette-Guerin vaccine against tuberculosis, a disease caused by Mycobacterium tuberculosis) have been show to reprogram the immune system, leading to enhanced protection against infection with disease-causing microorganisms unrelated to M. tuberculosis.

In this study, we will test the hypothesis that rabies vaccine has non-specific protective effects against common infectious disease (CID) syndromes (upper respiratory illness, diarrhea and fever) in a population of veterinary students. We will randomly assign previously-unvaccinated students who volunteer for the study to receive a primary course of three injections of rabies vaccine (experimental group) or an identical course of three injections of sterile water (control group). Participants will not know to which group they have been assigned. We will ask all participants to report episodes of illness through an online survey each week for 26 weeks, and will also record all clinically- and laboratory-confirmed cases of illness with CID syndromes. We hypothesize that rates of self-reported new episodes of CID illness over 26 weeks will be at least 25% lower in the experimental group, relative to the control group.

ELIGIBILITY:
Inclusion Criteria:

A student registered at RUSVM, and in the Veterinary Preparatory (VP) program or the 1st or 5th semester of the Doctor of Veterinary Medicine (DVM) program

Exclusion Criteria:

A student registered at RUSVM and in the VP program or the 1st or 5th semester of the DVM program will be excluded from the study if s/he:

1. has previously received a dose of rabies vaccine, or
2. is intending to undertake activities during the course of participation in the study that would increase their risk category of rabies exposure above that of the U.S. population at large, as defined by the Advisory Committee on Immunization Practices (ACIP) for human rabies prevention, or
3. does not provide informed consent for participation, or
4. enrolls in the study but does not present for the first injection within the first 12 weeks of the semester (up to and including Week 12), or
5. has a contraindication to rabies vaccine as described in the Rabivax-S package insert

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 546 (Actual)
Dates: Start 2018-08-29 (Actual); Primary Completion 2020-07-27 (Actual); Study Completion 2020-07-27 (Actual)

PRIMARY OUTCOMES:
Number of self-reported new episodes of acute common infectious disease (CID), defined as any of the following: upper respiratory illness (URI) or influenza-like illness (ILI) or diarrhea (DIA) or undifferentiated febrile illness (UFI) | Weekly self-reporting of occurrence or non-occurrence of episodes of CID for a maximum of 26 weeks, starting one week after allocation
  URI is defined as (two or more of the following: runny or blocked nose/sneezing/sore throat/cough) and (absence of itchy or watery eyes).
  ILI is defined as [fever (feeling feverish, or an axillary, oral or otic temperature of 100°F or higher)] and (cough or sore throat).
  DIA is defined as three or more loose stools within a 24-hour period.
  UFI is defined as [fever (feeling feverish, or an axillary, oral or otic temperature of 100°F or higher)] and (not meeting the case definition of URI, ILI or DIA).
  To be defined as a new episode, illness must be preceded by at least one week without any CID.

SECONDARY OUTCOMES:
Number of self-reported new episodes of respiratory illness (URI or ILI), DIA and UFI | Weekly self-reporting of occurrence or non-occurrence of episodes of respiratory illness, DIA and UFI for a maximum of 26 weeks, starting one week after allocation
Number of self-reported new weekly episodes of URI | Weekly self-reporting of occurrence or non-occurrence of episodes of URI for a maximum of 26 weeks, starting one week after allocation
  To be defined as a new episode, illness must be preceded by at least one week without any URI.
Number of self-reported new weekly episodes of ILI | Weekly self-reporting of occurrence or non-occurrence of episodes of ILI for a maximum of 26 weeks, starting one week after allocation
  To be defined as a new episode, illness must be preceded by at least one week without any ILI.
Number of self-reported new weekly episodes of DIA | Weekly self-reporting of occurrence or non-occurrence of episodes of DIA for a maximum of 26 weeks, starting one week after allocation
  To be defined as a new episode, illness must be preceded by at least one week without any DIA.
Number of self-reported new weekly episodes of UFI | Weekly self-reporting of occurrence or non-occurrence of episodes of UFI for a maximum of 26 weeks, starting one week after allocation
  To be defined as a new episode, illness must be preceded by at least one week without any UFI.
Number of clinically-confirmed episodes of CID syndromes | 27 weeks after allocation
  Clinically-confirmed episodes of CID syndromes, defined as an episode resulting in a visit to the RUSVM Student Health Services with a recorded ICD10 of J00 (acute nasopharyngitis); J11 (influenza due to unidentified influenza virus); R19.7 (diarrhea) or R50.9 (fever, unspecified).
Number of laboratory-confirmed episodes of CID syndromes | 27 weeks after allocation
  Laboratory-confirmed episodes of CID syndromes, defined as clinically-confirmed episodes with laboratory diagnosis of influenza virus, respiratory syncytial virus or metapneumovirus (URI/ILI episodes) or rotavirus or norovirus (DIA episodes)

CONTACTS AND LOCATIONS:
Overall Officials: Darryn Knobel, PhD, Principal Investigator — Ross University School of Veterinary Medicine
Locations (1):
- Ross University School of Veterinary Medicine, Basseterre, Saint Kitts and Nevis

REFERENCES:
- [Derived] Odita CI, Conan A, Smith-Antony M, Battice J, England S, Barry D, Gessner BD, Knobel DL. Non-specific effects of rabies vaccine on the incidence of self-reported common infectious disease episodes: A randomized controlled trial. Vaccine. 2022 Mar 8;40(11):1617-1623. doi: 10.1016/j.vaccine.2021.06.007. Epub 2021 Jun 11. PMID 34127294
- [Derived] Knobel D, Odita CI, Conan A, Barry D, Smith-Anthony M, Battice J, England S, Gessner BD. Non-specific effects of rabies vaccine on the incidence of common infectious disease episodes: study protocol for a randomized controlled trial. Trials. 2020 Jun 16;21(1):534. doi: 10.1186/s13063-020-04467-z. PMID 32546199

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-29): https://cdn.clinicaltrials.gov/large-docs/98/NCT03656198/Prot_SAP_000.pdf